CLINICAL TRIAL: NCT02526030
Title: Phase IV Study of Effectiveness of Aripiprazole, Quetiapine, and Ziprasidone in the Treatment of First Episode of Non-affective Psychosis Individuals Included in the First Episode Psychosis Clinical Program II (PAFIP II): a 3-year Follow-up
Brief Title: Comparative Study of Aripiprazole, Quetiapine and Ziprasidone in Treatment of First Episode Psychosis: 3-year Follow-up
Acronym: PAFIP2_3Y
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Marques de Valdecilla (Other)
Collaborators: Centro de Investigación Biomédica en Red de Salud Mental (Network); Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Benedicto Crespo-Facorro, Associate Professor of Psychiatry, Fundación Marques de Valdecilla
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZQ2005_3Y; CI 2005-0308007 (Other Grant/Funding Number: SENY Fundació Research Grant CI 2005-0308007)
Record Dates: First submitted 2015-08-12; First posted 2015-08-18 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Psychotic Disorders
Keywords: psychosis; antipsychotic agents; treatment; effectiveness
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Aripiprazole; Quetiapine Fumarate; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aripiprazole (Active Comparator): Oral, dose range 10-30 mg/day, once or twice a day, during study duration
  Interventions: Drug: Aripiprazole
- Quetiapine (Active Comparator): Oral, dose range 100-600 mg/day, once or twice a day, during study duration
  Interventions: Drug: Quetiapine
- Ziprasidone (Active Comparator): Oral, dose range 40-160 mg/day, once or twice a day, during study duration
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: Aripiprazole
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Quetiapine
  Other Names: Seroquel
  Arms: Quetiapine
Drug: Ziprasidone
  Other Names: Zeldox
  Arms: Ziprasidone

SUMMARY:
The selection of antipsychotic in early stages of the illness is mainly determined by its clinical effectiveness. Second generation antipsychotics (SGAs) are the first line drug treatment for individuals suffering from schizophrenia. It is clear that SGAs are not a homogeneous group and clinical effects and profile of side effects differ between SGAs. Differences among antipsychotics in terms of effectiveness have turned out to be a topic of increasing research interest, although comparisons between the different SGAs are scarce. In first episode of psychosis, SGAs have shown a higher treatment effectiveness compared to first generation antipsychotics (FGAs) (findings primarily driven by Haloperidol). Less evident seems to be the notion that some of the SGAs might be more effective (in terms of treatment discontinuation) than others. Most of the medium-term randomized studies have shown similar rates of all-cause treatment discontinuation in first episode patients treated with different SGAs. It may be concluded that more randomized controlled trails should be accomplished to determine the position of frequently used SGAs in clinical practice. Investigators undertook this study with the major objective of comparing the clinical effectiveness of three widely utilized SGAs (Aripiprazole, Ziprasidone and Quetiapine) in the acute treatment of first-episode non-affective psychosis individuals at 3 years of follow-up.

DETAILED DESCRIPTION:
Study setting and financial support: data for the present investigation were obtained from an ongoing epidemiological and three-year longitudinal intervention program of first-episode psychosis (PAFIP) conducted at the outpatient clinic and the inpatient unit at the University Hospital Marqués de Valdecilla, Spain. Conforming to international standards for research ethics, this program was approved by the local institutional review board. Patients meeting inclusion criteria and their families provided written informed consent to be included in the PAFIP. The Mental Health Services of Cantabria provided funding for implementing the program. None pharmaceutical company supplied any financial support to it.

Study design: the severity scale of the Clinical Global Impression (CGI) scale, the Brief Psychiatric Rating Scale (BPRS), the Scale for the Assessment of Positive symptoms (SAPS) and the Scale for the Assessment of Negative symptoms (SANS) were used to evaluate symptomatology. To assess general adverse event experiences the Scale of the Udvalg for Kliniske Undersogelser (UKU), the Simpson-Angus Rating Scale (SARS) and the Barnes Akathisia Scale (BAS) were used to assess side effects. The adverse events were evaluated using the UKU Side effect rating scale. Those treatment-emergent adverse events that occurred at a rate of at least 10% in either treatment group are considered. Treatment-emergent akathisia (BAS) and extrapyramidal symptoms (SARS) were assessed by both baseline-to-end changes and newly emergent categorical changes. The same trained psychiatrist (BC-F) completed all clinical assessments.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed in the First Episode Psychosis Clinical Program (PAFIP II) from October 2005 to January 2011.

Exclusion Criteria:

* Meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria for drug dependence
* Meeting DSM-IV criteria for mental retardation
* Having a history of neurological disease or head injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Effectiveness of antipsychotics (percentage of discontinuation of the initially assigned treatment) | 3 years
  Two measures for evaluate the effectiveness of antipsychotics:
  * Percentage of discontinuation of the initially assigned treatment: patients who completed the 3 years follow-up assessment and changed initial antipsychotic.
  * Mean time to all-cause medication discontinuation.
  Four reasons for the discontinuation were recorded: 1.- insufficient efficacy; 2.- marked side-effects; 3.- patient reported non-adherence and 4.- other causes. If more than one reason for discontinuation was present, the most important reason according to the above ranking was selected. Antipsychotic treatment data (doses, discontinuation and concomitant medications) were registered every 6 months. Insufficient efficacy was established at the treating physician's judgment only after at least three weeks of treatment.

SECONDARY OUTCOMES:
Change in general psychopathology measured by the Brief Psychiatric Rating Scale (BPRS) | 3 years
  Measured by BPRS.
Change in positive and negative symptoms measured by the Scale for the Assessment of Negative and Positive Symptoms (SANS and SAPS) | 3 years
  Measured by SANS and SAPS.
Adherence to treatment measured by Morinsky questionnaire | 3 years
  Adherence criteria for categorizing "good adherence category" using a 90% adherence as the cut-off will be set up as well based of infora. At study design we opted to set up stringent definition of "good adherence" because we were interested in differentiating individuals who really were good adherent and those with irregular taking to thoroughly investigate the impact of medication in illness outcome and biological parameters. Our results seem to point out the relevance of ensuring a good adherence (taking >90 % of prescribed medication) in early phases of the illness. Adherence to antipsychotic drugs was assessed by the information obtained from patients and close relatives by the staff (nurse, social worker and psychiatrists) involved in the clinical follow-up.
Functional outcome measured by Disability Assessment Scale (DAS) and Global Assessment Functioning (GAF). | 3 years
  DAS scores range from 0 (good social functioning) to 5 (bad social functioning). GAF scores range from 1 (many disease symptoms) to 100 (no disease symptoms).

OTHER OUTCOMES:
Relapse rate | 3 years
  Among patients who achieved clinical improvement and stability (CGI rating ≤ 4 and a decrease of at least 30% on BPRS total score and all BPRS key symptom items, by being rated ≤ 3 for more than 4 consecutive weeks at some point during the first 6 months following program entry), relapse was defined as any of the following criteria that occurred during follow-up: 1 - a rating of either 5 or above on any key BPRS symptom items, 2 - CGI rating of ≥ 6 and a change score of CGI of "much worse" or "very much worse", 3 - hospitalization for psychotic psychopathology, or 4 - completed suicide. The key BPRS symptoms were unusual thought content, hallucinations, suspiciousness, conceptual disorganization and bizarre behaviour. Exacerbation was defined as any 2-point increase of any of the key BPRS symptoms, excluding changes in which the rating remained at the non-psychotic level (i.e., <3).
Remission rate | 3 years
  Remission was defined according to Andreasen et al. (2005) criteria covering BPRS and SANS scores: 1.- a score of mild or less (≤3) on six predefined BPRS symptom items: grandiosity, suspiciousness, unusual thought content, hallucinations, conceptual disorganization and mannerisms; and 2.- SANS items scores of ≤2 simultaneously in all items. These criteria are required to be maintained for at least 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Benedicto Crespo-Facorro, Professor, Principal Investigator — University Hospital Marqués de Valdecilla, IDIVAL, Department of Psychiatry, School of Medicine, University of Cantabria, CIBERSAM Centro Investigación Biomédica en Red Salud Mental, Santander, Spain.
Locations (1):
- University Hospital Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez-Revuelta M, Pelayo-Teran JM, Juncal-Ruiz M, Vazquez-Bourgon J, Suarez-Pinilla P, Romero-Jimenez R, Setien Suero E, Ayesa-Arriola R, Crespo-Facorro B. Antipsychotic Treatment Effectiveness in First Episode of Psychosis: PAFIP 3-Year Follow-Up Randomized Clinical Trials Comparing Haloperidol, Olanzapine, Risperidone, Aripiprazole, Quetiapine, and Ziprasidone. Int J Neuropsychopharmacol. 2020 Apr 23;23(4):217-229. doi: 10.1093/ijnp/pyaa004. PMID 31974576
- [Derived] Gomez-Revuelta M, Pelayo-Teran JM, Juncal-Ruiz M, Ortiz-Garcia de la Foz V, Vazquez-Bourgon J, Gonzalez-Pinto A, Crespo-Facorro B. Long-Term Antipsychotic Effectiveness in First Episode of Psychosis: A 3-Year Follow-Up Randomized Clinical Trial Comparing Aripiprazole, Quetiapine, and Ziprasidone. Int J Neuropsychopharmacol. 2018 Dec 1;21(12):1090-1101. doi: 10.1093/ijnp/pyy082. PMID 30215723